CLINICAL TRIAL: NCT00914667
Title: An Open-Label, Randomized, Two-Way Crossover Study To Evaluate The Steady-State Effect Of Fesoterodine On The Pharmacokinetics And Pharmacodynamics Of A Single Supratherapeutic Dose Of Warfarin In Healthy Subjects.
Brief Title: The Effect Of Fesoterodine On Pharmacokinetics And Pharmacodynamics Of Warfarin In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A0221079
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder Urgency Frequency
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Warfarin; fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin Alone (Experimental): Reference treatment
  Interventions: Drug: warfarin
- Warfarin Concomitantly With Fesoterodine (Experimental): Test treatment
  Interventions: Drug: Warfarin plus Fesoterodine

INTERVENTIONS:
Drug: warfarin — Single Dose Warfarin 25 mg on Day 1
  Arms: Warfarin Alone
Drug: Warfarin plus Fesoterodine — Fesoterodine 8 mg ER tablets QD for 9 Days and Single Dose Warfarin 25 mg on Day 3
  Arms: Warfarin Concomitantly With Fesoterodine

SUMMARY:
This is an open-label, randomized, two-way crossover study to evaluate the steady-state effect of fesoterodine (8 mg QD) on the pharmacodynamics and pharmacokinetics of a single supratherapeutic dose of warfarin (25 mg) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years

Exclusion Criteria:

* Not healthy subjects--subjects with acute or chronic medical or psychiatric conditions or laboratory abnormality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Cmax and AUCinf for both S- and R-warfarin | 8 days per period
AUC_INR and INRmax | 8 days per period

SECONDARY OUTCOMES:
AUClast, Tmax and t½ for both S- and R-warfarin | 8 days per period
AUC_PT and PTmax | 8 days per period
Safety will be assessed by subjective symptoms/objective findings including physical examinations, clinical safety laboratory assessments, 12-lead ECGs, vital sign measurements and adverse event monitoring. | 8 days per period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221079&StudyName=The%20Effect%20Of%20Fesoterodine%20On%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Warfarin%20In%20Healthy%20Subjects